CLINICAL TRIAL: NCT00294190
Title: A Phase II Study Of Higher Dose Weekly Topotecan In The Treatment Of Patients With Extensive Stage Small-Cell Lung Cancer
Brief Title: Higher Dose Weekly Topotecan In The Treatment Of Patients With Extensive Stage Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 120; 105642
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2011-05

CONDITIONS: Small Cell Lung Cancer; Carcinoma, Small Cell
Keywords: Lung Cancer; Extensive stage; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Small Cell; Lung Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topotecan (Experimental)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — Topotecan 6mg/m2 IV weekly x 6 consecutive weeks followed by a 2 week break.
  Other Names: Hycamtin

SUMMARY:
This proposed phase II trial will investigate weekly topotecan at a higher dose than was used in the previous trials in an attempt to achieve improved response rates and disease control without added toxicity. To help ameliorate the fatigue, planned rest weeks will be incorporated into the schedule. This trial will be the first clinical trial to evaluate a higher dose of weekly topotecan in the treatment of extensive-stage SCLC.

DETAILED DESCRIPTION:
All patients will receive weekly topotecan.

Topotecan 6mg/m2 IV weekly x 6 consecutive weeks followed by a 2 week break. Cycles are repeated every 8 weeks, for 3 cycles. Restaging studies will be performed every cycle (or 8 weeks.)

ELIGIBILITY:
Inclusion Criteria:

* Extensive small cell lung cancer with progression after one previous chemotherapy or chemotherapy/radiation therapy regimen
* Measurable or evaluable disease
* Able to perform activities of daily living with minimal assistance
* Adequate bone marrow, liver and kidney function
* May have received no more than 3 previous courses of radiation therapy
* Give written informed consent prior to study entry

Exclusion Criteria:

* Patients with limited stage disease
* History of a prior malignancy within three years
* Female patients who are pregnant or are breast feeding
* Significant history of uncontrolled cardiac disease
* Myocardial infarction or stroke within six months
* Symptomatic peripheral vascular disease
* CNS involvement
* Serious active infection or underlying medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 18 months

SECONDARY OUTCOMES:
overall toxicity | 18 months
time to progression | 18 months
duration of response | 18 months
overall survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Derived] Spigel DR, Greco FA, Burris HA 3rd, Shipley DL, Clark BL, Whorf RC, Arrowsmith ER, Hainsworth JD. A phase II study of higher dose weekly topotecan in relapsed small-cell lung cancer. Clin Lung Cancer. 2011 May;12(3):187-91. doi: 10.1016/j.cllc.2011.03.016. Epub 2011 Apr 28. PMID 21663862